CLINICAL TRIAL: NCT02449213
Title: A Biobehavioral Model of Diabetes Risk in Chinese Immigrants
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-8006
Record Dates: First submitted 2015-05-17; First posted 2015-05-20 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, and hair samples will be obtained
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, longitudinal study of Chinese American immigrants will examine whether psychosocial factors (e.g., acculturative stress, social isolation, discrimination) are associated with markers of type 2 diabetes risk over time, and whether such associations are mediated by inflammatory pathways.

DETAILED DESCRIPTION:
It is now well-documented that immigration to the US leads to increased risk for various chronic diseases, including type 2 diabetes. The increased diabetes risk observed among Chinese immigrants has been primarily attributed to changes in diet and weight gain following immigration, but these changes can only partially explain disparities in disease risk. Models of immigrant health suggest that the stress of adapting to life in a new country has a considerable impact on physical health. However, few studies have considered the psychosocial impact of immigration upon biomarkers of health and disease risk. Therefore, this longitudinal study of US Chinese immigrant men and women will examine: (1) whether psychosocial factors (e.g., acculturative stress, social isolation, discrimination) are associated with markers of type 2 diabetes risk over time; and (2) whether the association between psychosocial factors and diabetes risk markers is mediated by inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Chinese heritage;
* migration from Asia in adulthood (aged 18 years or older); and
* age 35-65 years

Exclusion Criteria:

* Current or prior history of diabetes
* Self-reported conditions of cancer, auto-immune disorders, HIV, or psychiatric illness
* Use of medications that may impact study outcomes (e.g., steroidal or non-steroidal anti-inflammatory medications)
* Inability to provide informed consent.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 600 foreign-born Chinese Americans
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 24 months post-baseline
  Insulin resistance will be estimated according to the homeostasis model assessment (HOMA) as HOMA = (fasting insulin x fasting glucose) / 22.5

SECONDARY OUTCOMES:
glycated hemoglobin (HbA1c) | 24-months post-baseline
  Level of blood sugar

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y. Fang, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States